CLINICAL TRIAL: NCT01144052
Title: De-escalation After Natalizumab Treatment With Interferon-beta-1b in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Natalizumab De-escalation With Interferon Beta-1b
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Claudio Gobbi (Other Government)
Collaborators: Ospedale Civico, Lugano (Other Government)
Responsible Party: Sponsor-Investigator, Claudio Gobbi, Dr. med., Ospedale Civico, Lugano
Organization: Ospedale Civico, Lugano (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EOC.NC.09.01
Record Dates: First submitted 2010-06-11; First posted 2010-06-15 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Natalizumab; Interferon-beta 1b; De-escalation; Ticino
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b; Natalizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Natalizumab (Active Comparator): Eligible patients to this study have been treated with monthly infusions of natalizumab for at least 12 months at study entry. Natalizumab continues to be administered every four weeks by intravenous infusion from the beginning of the study as indicated by the manufacturers' instructions.
  Interventions: Drug: Natalizumab
- Interferon-beta-1b (Experimental): 250 mcg (8 MIU) subcutaneous injections every other day
  Interventions: Drug: interferon beta-1b

INTERVENTIONS:
Drug: interferon beta-1b — Eligible patients to this study have been treated with monthly infusions of natalizumab for at least 12 month at study entry. After a wash-out period of one month, interferon-beta-1b will be administered subcutaneously every other day as indicated by the manufacturers' instructions including the stepwise up-titration scheme as recommended for treatment start. The final dose of interferon beta-1b is 250 mcg (8 million International Units [MIU])
  Other Names: Betaferon®
  Arms: Interferon-beta-1b
Drug: Natalizumab — Eligible patients to this study have been treated with monthly infusions of natalizumab for at least 12 months at study entry. Natalizumab continues to be administered every four weeks by intravenous infusion from the beginning of the study as indicated by the manufacturers' instructions.
  Other Names: Tysabri
  Arms: Natalizumab

SUMMARY:
Multiple Sclerosis (MS) is the most common neurological disorder causing disability in young adults. The management of MS-patients requires treatment with disease-modifying agents, monoclonal antibodies such as natalizumab or immunosuppressants. Natalizumab showed good efficacy and is approved for treatment of relapsing MS with a number of restrictions due to safety issues. Cognitive data related to natalizumab treatment are still scarce. Interferon-beta-1b is approved for high-frequency, subcutaneous (sc) administration in the treatment of multiple sclerosis. It reduces the relapse rate, severity, hospitalisation and the disease activity as seen on MRI.

This is a pilot study to explore the concept of de-escalating natalizumab treatment to interferon-beta-1b e.o.d compared to continuous treatment with natalizumab in patients with relapsing-remitting multiple sclerosis previously treated with natalizumab for 12 months. The study is designed as prospective, controlled, randomized, rater-blinded, parallel-group, two arm, mono-centric including patients of the Ticino Cohort. One arm will be treated with Interferon-beta 1b 250mcg given subcutaneously every other day, the other with Natalizumab 300 mg given intravenously (i.v.), every four weeks. The treatment duration is 12 months, the follow-up period 12 months. The time to first on-study relapse will be compared between the to treatment arms (primary outcome). Other efficacy parameter include clinical and radiological parameters, patient reported outcome on quality of life and fatigue. Safety is assessed by reports of adverse events.

DETAILED DESCRIPTION:
At present, there is no cure for multiple sclerosis and the management of MS-patients requires treatment with disease-modifying agents such as interferon-beta or glatiramer acetate, monoclonal antibodies such as natalizumab or immunsuppressants such as mitoxantrone, azathioprine or methotrexate. Acute relapses are usually treated with corticosteroids. Natalizumab is a humanized monoclonal antibody directed against α4-integrin, a component of VLA-4 (very late antigen-4) present on leukocytes. Following submission of additional safety data, the agencies such as Swissmedic or EMEA have issued approval of natalizumab for treatment of relapsing MS with a number of restrictions. The preparation has been available in Switzerland since 2006. According to the current scientific information, natalizumab (Tysabri®) is indicated as a "disease-modifying monotherapy of highly active relapsing MS" for the following patient groups: 1) patients showing high levels of disease activity despite treatment with an IFN-β preparation, or 2) untreated/treatment-naive patients with rapidly progressing relapsing-remitting MS (at least two serious relapses per year).

The primary objective of this pilot study is to generate first data and hypotheses on the concept of de-escalating natalizumab-treated relapsing-remitting multiple sclerosis patients to interferon-beta-1b e.o.d compared to continuous treatment on natalizumab for planning of further clinical studies regarding safety and efficacy.

As secondary objectives, clinical, neuropsychological parameters, MRI and laboratory parameter and safety aspects will be assessed in accordance to the protocol available for the management of patient on natalizumab at our service.

This is a prospective, controlled, randomized, rater-blinded, parallel-group, monocentric, two arm, phase IV pilot study. Patients with relapsing-remitting forms of MS, respecting all inclusion/exclusion criteria, will be randomized into two equal-size parallel arms for de-escalation to interferon beta-1b (after a month wash-out) or for continued treatment on natalizumab.

it is planned to enrol 20 patients (1/2 in the natalizumab group, 1/2 in the interferon beta-1b group. Patients providing written informed consent will be treated for 12 months; pre-planned follow-up of further 12 month

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients with relapsing-remitting forms of multiple sclerosis (according to McDonald's criteria)
* Age between 18 and 60 years
* Natalizumab-treatment for at least 12 month following the current Swiss guidelines for treatment initiation
* Eligible patients are clinically stable (free from relapses and 6-month confirmed disability progression for at least 6 months) while on natalizumab-treatment
* Women of potential childbearing with active contraceptive methods
* Patients who are willing to undergo study procedures
* Patients who are willing and able to sign informed consent

Exclusion Criteria:

* Patients who have previously entered this study
* Natalizumab-treatment for less than 12 month following the current Swiss guidelines for treatment initiation
* Sign of clinical disease activity within the 6 month
* One or more relapses and/or 6-month confirmed disability progression during the 6 months prior to the study
* Any disease other than multiple sclerosis that would better explain the patient's signs and symptoms
* Secondary progressive MS
* Primary progressive MS
* Pregnancy - Urine pregnancy test at baseline visit - or breast feeding
* Uncontrolled, clinically significant heart diseases, such as arrhythmias, angina, or uncompensated congestive heart failure
* History of severe depression or attempted suicide or current suicidal ideation
* Medical or psychiatric conditions that compromise the ability to give informed consent, to comply with the protocol, or to complete the study
* Uncontrolled seizure disorder
* Myopathy or clinically significant liver disease
* Inability, in the opinion of the principal investigator or staff, to comply with protocol requirements for the duration of the study
* Known hypersensitivity to interferon-beta or other human proteins including albumin
* Any contraindication for MRI or contrast administration
* A history of drug abuse in the 6 months prior to screening
* Treatment with any of the following in the 30 days before day 1: systemic corticosteroids, ACTH, or other investigational drugs.
* Participation in any other study involving investigational or marketed products, concomitantly or within 30 days prior to entry in the study
* Current participation on other clinical trials
* Treatment with drugs which might interfere with the evaluation of study drugs during the study protocol
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Gobbi, Dr med., Principal Investigator — Neurocenter of Southern Switzerland, Ospedale Civico Lugano
Locations (1):
- Neurocenter of Southern Switzerland, Ospedale Civico Lugano, Lugano, Canton Ticino, Switzerland

REFERENCES:
- [Background] Multiple Sclerosis Therapy Consensus Group (MSTCG); Wiendl H, Toyka KV, Rieckmann P, Gold R, Hartung HP, Hohlfeld R. Basic and escalating immunomodulatory treatments in multiple sclerosis: current therapeutic recommendations. J Neurol. 2008 Oct;255(10):1449-63. doi: 10.1007/s00415-008-0061-1. Epub 2008 Oct 29. PMID 19005625
- [Background] Rudick RA, Stuart WH, Calabresi PA, Confavreux C, Galetta SL, Radue EW, Lublin FD, Weinstock-Guttman B, Wynn DR, Lynn F, Panzara MA, Sandrock AW; SENTINEL Investigators. Natalizumab plus interferon beta-1a for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):911-23. doi: 10.1056/NEJMoa044396. PMID 16510745
- [Background] Polman CH, O'Connor PW, Havrdova E, Hutchinson M, Kappos L, Miller DH, Phillips JT, Lublin FD, Giovannoni G, Wajgt A, Toal M, Lynn F, Panzara MA, Sandrock AW; AFFIRM Investigators. A randomized, placebo-controlled trial of natalizumab for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):899-910. doi: 10.1056/NEJMoa044397. PMID 16510744
- [Background] IFNB Multiple Sclerosis Study Group. Interferon beta-lb is effective in relapsing-remitting multiple sclerosis. I. Clinical results of a multicenter, randomized, double-blind, placebo-controlled trial. 1993 [classical article]. Neurology. 2001 Dec;57(12 Suppl 5):S3-9. No abstract available. PMID 11902592
- [Background] Paty DW, Li DK; UBC MS/MRI Study Group and IFNB Multiple Sclerosis Study Group. Interferon beta-lb is effective in relapsing-remitting multiple sclerosis. II. MRI analysis results of a multicenter, randomized, double-blind, placebo-controlled trial. 1993 [classical article]. Neurology. 2001 Dec;57(12 Suppl 5):S10-5. No abstract available. PMID 11902589
- [Background] Putzki N, Yaldizli O, Tettenborn B, Diener HC. Multiple sclerosis associated fatigue during natalizumab treatment. J Neurol Sci. 2009 Oct 15;285(1-2):109-13. doi: 10.1016/j.jns.2009.06.004. Epub 2009 Jun 26. PMID 19560168
- [Background] Ransohoff RM. Natalizumab and PML. Nat Neurosci. 2005 Oct;8(10):1275. doi: 10.1038/nn1005-1275. No abstract available. PMID 16189528
- [Background] Sadovnick AD, Ebers GC. Epidemiology of multiple sclerosis: a critical overview. Can J Neurol Sci. 1993 Feb;20(1):17-29. doi: 10.1017/s0317167100047351. PMID 8467424
- [Result] Gobbi C, Meier DS, Cotton F, Sintzel M, Leppert D, Guttmann CR, Zecca C. Interferon beta 1b following natalizumab discontinuation: one year, randomized, prospective, pilot trial. BMC Neurol. 2013 Aug 2;13:101. doi: 10.1186/1471-2377-13-101. PMID 23915113
- [Result] Zecca C, Riccitelli GC, Calabrese P, Pravata E, Candrian U, Guttmann CR, Gobbi C. Treatment satisfaction, adherence and behavioral assessment in patients de-escalating from natalizumab to interferon beta. BMC Neurol. 2014 Feb 28;14:38. doi: 10.1186/1471-2377-14-38. PMID 24576156
- See also: Homepage of the hospital organisation in Ticino — http://www.eoc.ch
- See also: Homepage of the Swiss Society of Multiple Sclerosis — http://www.multiplesklerose.ch

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 2010 to 2011 Out-patients of Neurology ambulatory
Period: Overall Study
Arm/Group | Natalizumab | Interferon-beta-1b
Started | 10 | 9
Completed | 9 | 8
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Natalizumab | Interferon-beta-1b | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (10.83) | 39 (13.26) | 41 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  Switzerland | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Until First On-study Relapse
Description: Patients were followed-up during 12 months and time to first on-study relapse from randomization was recorded.
Time Frame: 12 months
Population: All enrolled and randomized patients fulfilled the criteria for analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Natalizumab | Interferon-beta-1b
Number analyzed (Participants) | 10 | 9
days | NA [NA to NA] — This value is not available, because zero patients experienced a relapse. | 103 [103 to 103]
Statistical Analysis 1: Comparison: Natalizumab vs Interferon-beta-1b; Test type: Non-Inferiority or Equivalence — No statistical hypothesis tests for efficacy were performed as this was a pilot study serving to generate first data and hypotheses; p = 0.125, Log Rank

2. Secondary Outcome: Number of Participants With Relapses
Time Frame: 12 months
Population: All enrolled and randomized patients were analyzed.
Measure: Number; unit: participants
Arm/Group | Natalizumab | Interferon-beta-1b
Number analyzed (Participants) | 10 | 9
participants | 0 | 2
Statistical Analysis 1: Comparison: Natalizumab vs Interferon-beta-1b; Test type: Superiority or Other; p = 0.447, non-parametric

3. Secondary Outcome: Number of Relapses
Time Frame: 12 months
Measure: Number; unit: number of events
Arm/Group | Natalizumab | Interferon-beta-1b
Number analyzed (Participants) | 10 | 9
number of events | 0 | 3
Statistical Analysis 1: Comparison: Natalizumab vs Interferon-beta-1b; Test type: Superiority or Other; p = 0.447, non-parametric

4. Secondary Outcome: Proportion of Relapse Free Patients
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Natalizumab | Interferon-beta-1b
Number analyzed (Participants) | 10 | 9
participants | 10 | 7
Statistical Analysis 1: Comparison: Natalizumab vs Interferon-beta-1b; Test type: Superiority or Other; p = 0.206, t-test, 2 sided

5. Secondary Outcome: Severity of Relapses
Description: Change of Expanded Disability Status Scale (EDSS 1-10). Higher values represent a worser outcome.
Time Frame: 12 months vs baseline
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Natalizumab | Interferon-beta-1b
Number analyzed (Participants) | 10 | 9
units on a scale | 0 [0 to 0] | 0.5 [0.5 to 1.5]

6. Secondary Outcome: MRI Parameters
Description: Number of new T2-hyperintense lesions, Number of Gd-enhancing lesions on T1-weighted images. Assessments at month 3, 6, 9, 12, 18, 24.
Time Frame: 12 months
Population: All enrolled and randomized patients were analyzed.
Measure: Median (Full Range); unit: Lesions
Arm/Group | Natalizumab | Interferon-beta-1b
Number analyzed (Participants) | 10 | 9
Lesions
  nT2L month 3 | 0 [0 to 1] | 0.5 [0 to 2]
  nT2L month 6 | 0 [0 to 2] | 1.5 [0 to 9]
  nT2L month 9 | 0 [0 to 0] | 0.5 [0 to 6]
  nT2L month 12 | 0 [0 to 0] | 0 [0 to 12]
  GD+L month 3 | 0 [0 to 0] | 0 [0 to 1]
  GD+L month 6 | 0 [0 to 0] | 0 [0 to 5]
  GD+L month 9 | 0 [0 to 0] | 0 [0 to 1]
  GD+L month 12 | 0 [0 to 1] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Natalizumab vs Interferon-beta-1b; Test type: Non-Inferiority or Equivalence — No statistical hypothesis tests for efficacy were performed, as this was pilot study serving to generate first data and hypotheses; p = 0.234, Wilcoxon (Mann-Whitney); p-value refers to nT2L at month 12

7. Secondary Outcome: Number of Patients With Adverse Events
Description: Recording and reporting according to regulations. Monthly assessments or if necessary.
Time Frame: 12 months
Population: All patients enrolled and randomized were analyzed.
Measure: Number; unit: participants
Arm/Group | Natalizumab | Interferon-beta-1b
Number analyzed (Participants) | 10 | 9
participants
  Number of patients with infections | 7 | 4
  Number of patients with injections site reactions | 0 | 4

8. Secondary Outcome: Number of Infections
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | Natalizumab | Interferon-beta-1b
Number analyzed (Participants) | 10 | 9
events | 25 | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 12 months of the trial
Arm/Group | Natalizumab | Interferon-beta-1b
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/9
Other Adverse Events (participants affected / at risk) | 7/10 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natalizumab (N=10) | Interferon-beta-1b (N=9)
gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — One patient in the NTZ arm experienced a gastroenteritis requiring his hospitalisation. The patient recovered without sequelae and continued the study. The adverse event was judged to be unrelated to the study medication.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natalizumab (N=10) | Interferon-beta-1b (N=9)
Infection (Infections and infestations) | 7 (7) | 3 (3)
Injection site reaction (Investigations) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No